CLINICAL TRIAL: NCT04576780
Title: An Integrated Strategy for the Expedited Diagnosis, Referral, Assessment and Treatment of Complex Colorectal Polyps
Brief Title: An Integrated Management Pathway for Complex Colorectal Polyps
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: CTO - 1899
Record Dates: First submitted 2020-09-15; First posted 2020-10-06 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Polyp Colorectal
Keywords: Large Colorectal Polyp; Complex Colorectal Polyp

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Referred Patients with Large, Complex Colorectal Polyps: Patients referred from outside community care hospitals or ambulatory endoscopy centers to the therapeutic endoscopy group at St. Michaels Hospital via the new integrated management pathway for endoscopic resection of a large or complex colorectal polyp.
  Interventions: Other: Integrated Large Complex Polyp Referral Pathway

INTERVENTIONS:
Other: Integrated Large Complex Polyp Referral Pathway — The referring doctor will use a standardized template to send the referral along with its associated video or high-resolution photographs.
  Referrals will be reviewed in a consensus fashion by at least 2 expert physicians at St. Michael's Hospital (SMH) on a bi-weekly basis. Polyps will be scored using a standardized evaluation form that documents relevant polyp features to assist the determination of whether a lesion is amenable to curative endoscopic resection.
  Cases will be triaged as being: (1) a standard polyp suitable for local removal in the community; (2) a complex polyp requiring expert removal at SMH with priority assigned based on the suspected risk of invasive disease; (3) a polyp that is not amenable to endoscopic resection or that is suspicious for cancer will that be recommended for surgical resection.

SUMMARY:
The purpose of this study is to evaluate the impact of implementing an integrated clinical care pathway for the diagnosis, referral, evaluation and treatment of large complex colorectal polyps on clinical outcomes

DETAILED DESCRIPTION:
Our project will create a system that links community hospitals and ambulatory endoscopy centers throughout the province of Ontario, directly to the expert endoscopists at our tertiary referral center, to facilitate the timely assessment of polyps based on an electronic referral containing endoscopic video recordings or high-resolution images rather than a paper report through a centralized referral pathway. This polyp adjudication will happen in a timely fashion without involving in-person patient consultation, and will streamline the management of these patients to either referral for surgery or booking for endoscopic polyp removal by therapeutic colonoscopy at our center. Specific endoscopy time slots will be reserved for these patients to ensure they have efficient access to their treatment. This system represents a new care model for managing patients with concerning pre-cancerous lesions diagnosed in disparate local hospitals through a centralized process of referral, diagnostic evaluation and treatment at an expert tertiary referral centre.

The primary aim of our study will be to track the outcomes of the new standard-of-care clinical pathway. Clinical objectives of the project include a reduction in wait times for expert assessment after diagnosis of a large or otherwise concerning polyp combined with reduced wait times for therapeutic removal of these polyps, minimizing unnecessary surgery for benign lesions, and facilitating early recommendation for surgery in those patients who truly require surgical resection. Additional objectives include the achievement of excellent rates of clinical success, complication rates similar to those reported in the literature, and high levels of satisfaction from referring doctors at participating centers. A final, major goal is to assess whether this pilot program could serve as a model to be expanded to other academic, tertiary referral centers throughout the province of Ontario.

Our primary research question seeks to compare the diagnostic accuracy of expert polyp adjudication between the different modes of referral (video clip, color photograph, faxed images) against the real-time endoscopic diagnosis during therapeutic colonoscopy and the final pathologic result. The secondary research question is to follow the clinical outcomes of all patients who undergo endoscopic mucosal resection (EMR) of a large or complex colorectal polyp to evaluate the efficacy and safety of this procedure at our expert tertiary referral center.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient 18 years or older
* Large or complex colorectal polyp found during diagnostic colonoscopy

Exclusion Criteria:

* Severe medical comorbidities that contraindicate safe endoscopy procedures
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who were identified to have a large, complex polyp on colonoscopy at a community hospital or ambulatory endoscopy center referred for removal to the therapeutic endoscopy group at St. Michaels Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of remote polyp diagnosis (based on video clips, electronic color photographs or paper-based images) compared to real-time endoscopic diagnosis during therapeutic colonoscopy | During Procedure
  Determination of diagnostic accuracy (reported as sensitivity and specificity) of video-based vs. real-time endoscopic diagnosis of polyps; diagnostic accuracy of electronic color photo-based vs. real-time endoscopic diagnosis of polyps; diagnostic accuracy of paper-based images vs. real-time endoscopic diagnosis of polyps.

SECONDARY OUTCOMES:
Patient Wait Times | During Procedure
  Wait times (measured in days) from index colonoscopy to polyp adjudication, and from index colonoscopy to therapeutic polyp removal. Comparison will be made to historical wait times for polyps > 2 cm referred to SMH for polyp removal.
Prediction of Polyp Diagnosis | Until availability of histology, generally up to 2 weeks post procedure
  Polyp diagnosis based on initial colonoscopy performed at the referring centre, video- or photo-based assessment during polyp triage, and real-time evaluation during colonoscopy by expert endoscopist at SMH, assessed against final pathology from resected polyp specimen.
Need for adjunctive removal | During Procedure
  Rate of complete snare resection of polyps versus need for the use of combined adjunctive techniques (hot/cold avulsion, argon plasma coagulation, etc.) to achieve removal of polyps.
Prediction of Successful Endoscopic Treatment | Through study completion, up to 1 year
  Accuracy (reported as likelihood ratios) of the correct prediction of successful endoscopic treatment based on initial video-based, electronic colour photo-based, or paper image-based assessment during polyp triage compared to real-time evaluation during colonoscopy (prior to commencing attempt at polyp removal), assessed against final endoscopic outcome.
Procedural complications | Up to 4 weeks
  Rate of immediate and delayed complications both intra-procedural and post-procedural up to 4 weeks.
Residual/Recurrent Polyp | 6 months
  Rate and predictors of residual or recurrent polyp at follow-up surveillance colonoscopy.
Referring Physician Satisfaction | 1 year
  Study specific survey consisting of a 5 point likert scale ranging from 1 ("extremely dissatisfied") to 5 ("extremely satisfied"). Assessed at 1 year from initial referral.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Teshima, MD, Principal Investigator — St. Michaels Hospital

DOCUMENTS (1):
  • Informed Consent Form (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT04576780/ICF_000.pdf